CLINICAL TRIAL: NCT02277938
Title: Urinary Excretion of Acetylamantadine by Cancer Patients
Brief Title: Acetylamantadine Excretion by Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Collaborators: BioMark Technologies Inc. (Industry); St. Boniface Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2012:063
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Amantadine; Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — saliva, blood, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Amantadine: Lung cancer patients being prescribed chemotherapy
  Interventions: Drug: Amantadine

INTERVENTIONS:
Drug: Amantadine — Amantadine is a drug that has been on the market for several years and is currently approved for the treatment of Parkinson's disease and for prevention against influenza A infection. Amantadine may be of value in detecting the presence of cancer.
  Other Names: Systemic chemotherapy

SUMMARY:
Several factors discourage the implementation of cancer screening to the population in general, which would result in earlier diagnosis and an expected improved survival. Concurrent in vivo and in vitro research has shown that drug acetylation activity is increased in cancer. Amantadine may be of value in detecting the presence of cancer. Accordingly, this study will examine how Amantadine is eliminated by the body in cancer patients. This is an important step in validating a cancer detection method that can be implemented economically for screening of large numbers of people.

DETAILED DESCRIPTION:
The study will involve the screening of volunteer patients with various types of cancer to provide a first indication of which types of cancer and at what stage of tumor burden acetylamantadine will be found in patients' plasma, saliva and urine samples. Volunteers will provide complete first morning urine collection prior to amantadine ingestion. The volunteers will then ingest a therapeutic dose of amantadine (200 mg: 2x100mg capsules), at least 2 hours before breakfast (nothing to eat or drink except water after midnight before the scheduled appointment), and their complete urine will be collected at 2 and 4 hours (plus or minus 1 hour) after amantadine ingestion. In addition, blood samples will be taken by venipuncture before and at 2 and 4 hours after drug ingestion. The patients will be asked to provide a saliva sample at the same time as the urine samples are taken after drug ingestion.

ELIGIBILITY:
Inclusion Criteria: newly diagnosed or untreated cancer (GI, lung, prostate and breast cancer)

-

Exclusion Criteria: Any previous adverse reaction to Amantadine

* currently pregnant or lactating

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed cancer
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2013-08 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Acetylated Amantadine levels in urine | 2 and 4 hours after Amantadine ingestion
  Change in acetylamantadine excretion

CONTACTS AND LOCATIONS:
Locations (1):
- St. Boniface Hospital, Winnipeg, Manitoba, Canada

REFERENCES:
- [Result] Young RC. Cancer statistics, 2002: progress or cause for concern? CA Cancer J Clin. 2002 Jan-Feb;52(1):6-7. doi: 10.3322/canjclin.52.1.6. No abstract available. PMID 11814066
- [Result] Smith RA, Cokkinides V, von Eschenbach AC, Levin B, Cohen C, Runowicz CD, Sener S, Saslow D, Eyre HJ; American Cancer Society. American Cancer Society guidelines for the early detection of cancer. CA Cancer J Clin. 2002 Jan-Feb;52(1):8-22. doi: 10.3322/canjclin.52.1.8. PMID 11814067
- [Result] Bras AP, Hoff HR, Aoki FY, Sitar DS. Amantadine acetylation may be effected by acetyltransferases other than NAT1 or NAT2. Can J Physiol Pharmacol. 1998 Jul-Aug;76(7-8):701-6. doi: 10.1139/cjpp-76-7-8-701. PMID 10030449
- [Result] Bras AP, Janne J, Porter CW, Sitar DS. Spermidine/spermine n(1)-acetyltransferase catalyzes amantadine acetylation. Drug Metab Dispos. 2001 May;29(5):676-80. PMID 11302933
- [Result] Matsui I, Wiegand L, Pegg AE. Properties of spermidine N-acetyltransferase from livers of rats treated with carbon tetrachloride and its role in the conversion of spermidine into putrescine. J Biol Chem. 1981 Mar 10;256(5):2454-9. No abstract available. PMID 7007382
- [Result] Pegg AE, Seely JE, Poso H, della Ragione F, Zagon IA. Polyamine biosynthesis and interconversion in rodent tissues. Fed Proc. 1982 Dec;41(14):3065-72. PMID 7141002
- [Result] Seiler N. Functions of polyamine acetylation. Can J Physiol Pharmacol. 1987 Oct;65(10):2024-35. doi: 10.1139/y87-317. PMID 3322538
- [Result] Bettuzzi S, Davalli P, Astancolle S, Carani C, Madeo B, Tampieri A, Corti A. Tumor progression is accompanied by significant changes in the levels of expression of polyamine metabolism regulatory genes and clusterin (sulfated glycoprotein 2) in human prostate cancer specimens. Cancer Res. 2000 Jan 1;60(1):28-34. Erratum In: Cancer Res 2000 Mar 1;60(5):1472. Saverio, B [corrected to Bettuzzi, S]; Pierpaola, D [corrected to Davalli, P]; Serenella, A [corrected to Astancolle, S]; ,C [corrected to Carani, C]; Bruno, M [corrected to Madeo, B]; Auro, T [corrected to Tampieri, A]; Arnaldo, C [corrected to Corti, A]. PMID 10646846
- [Result] Russell DH. Increased polyamine concentrations in the urine of human cancer patients. Nat New Biol. 1971 Sep 29;233(39):144-5. doi: 10.1038/newbio233144a0. No abstract available. PMID 5286749
- [Result] Suh JW, Lee SH, Chung BC, Park J. Urinary polyamine evaluation for effective diagnosis of various cancers. J Chromatogr B Biomed Sci Appl. 1997 Jan 24;688(2):179-86. doi: 10.1016/s0378-4347(96)00266-6. PMID 9061454
- [Result] Takenoshita S, Matsuzaki S, Nakano G, Kimura H, Hoshi H, Shoda H, Nakamura T. Selective elevation of the N1-acetylspermidine level in human colorectal adenocarcinomas. Cancer Res. 1984 Feb;44(2):845-7. PMID 6692383
- [Result] Kingsnorth AN, Wallace HM. Elevation of monoacetylated polyamines in human breast cancers. Eur J Cancer Clin Oncol. 1985 Sep;21(9):1057-62. doi: 10.1016/0277-5379(85)90291-3. PMID 4065178
- [Result] Pine MJ, Huben RP, Pegg AE. Production of N1-acetyl spermidine by renal cell tumors. J Urol. 1989 Mar;141(3):651-5. doi: 10.1016/s0022-5347(17)40925-6. PMID 2493102
- [Result] Sessa A, Perin A. Increased synthesis of N1-acetylspermidine in hepatic preneoplastic nodules and hepatomas. Cancer Lett. 1991 Feb;56(2):159-63. doi: 10.1016/0304-3835(91)90091-u. PMID 1998945
- [Result] Dilman VM, Anisimov VN, Kolosov AI, Bulovskaya LN. On the relationship between the activity of acetylation, growth of experimental tumors and efficacy of their suppression by hydrazine sulphate. Oncology. 1976;33(5-6):219-21. doi: 10.1159/000225149. PMID 1026855
- [Result] Bulovskaya LN, Krupkin RG, Bochina TA, Shipkova AA, Pavlova MV. Acetylator phenotype in patients with breast cancer. Oncology. 1978;35(4):185-8. doi: 10.1159/000225282. PMID 704038
- [Result] Chekharina YeA, Bulovskaya LN, Pavlova MV, Krupkin RG. Activity of N-acetyltransferase in patients with malignant lymphomas. Neoplasma. 1978;25(4):471-5. PMID 692806
- [Result] Geylan YS, Dizbay S, Guray T. Arylamine N-acetyltransferase activities in human breast cancer tissues. Neoplasma. 2001;48(2):108-11. PMID 11478689
- [Result] Estrada-Rodgers L, Levy GN, Weber WW. Characterization of a hormone response element in the mouse N-acetyltransferase 2 (Nat2*) promoter. Gene Expr. 1998;7(1):13-24. PMID 9572394
- [Result] Olsen H, Morland J. Ethanol-induced increase in drug acetylation in man and isolated rat liver cells. Br Med J. 1978 Nov 4;2(6147):1260-2. doi: 10.1136/bmj.2.6147.1260. PMID 709306
- [Result] Olsen H, Morland J. Ethanol-induced increase in procainamide acetylation in man. Br J Clin Pharmacol. 1982 Feb;13(2):203-8. doi: 10.1111/j.1365-2125.1982.tb01357.x. PMID 7059417
- [Result] LESTER D. THE ACETYLATION OF ISONIAZID IN ALCOHOLICS. Q J Stud Alcohol. 1964 Sep;25:541-3. No abstract available. PMID 14211150
- [Result] Thomas BH, Solomonraj G. Drug interactions with isoniazid metabolism in rats. J Pharm Sci. 1977 Sep;66(9):1322-6. doi: 10.1002/jps.2600660930. PMID 903875
- [Result] Obayashi M, Matsui-Yuasa I, Kitano A, Kobayashi K, Otani S. Posttranslational regulation of spermidine/spermine N1-acetyltransferase with stress. Biochim Biophys Acta. 1992 May 7;1131(1):41-6. doi: 10.1016/0167-4781(92)90096-i. PMID 1581359
- [Result] Perin A, Sessa A. Polyamine acetylation in rat liver following long-term ethanol ingestion. Biochim Biophys Acta. 1993 Feb 13;1156(2):113-6. doi: 10.1016/0304-4165(93)90124-q. PMID 8427870
- [Result] Aoki FY, Sitar DS. Clinical pharmacokinetics of amantadine hydrochloride. Clin Pharmacokinet. 1988 Jan;14(1):35-51. doi: 10.2165/00003088-198814010-00003. PMID 3280212
- [Result] Gaudry SE, Sitar DS, Smyth DD, McKenzie JK, Aoki FY. Gender and age as factors in the inhibition of renal clearance of amantadine by quinine and quinidine. Clin Pharmacol Ther. 1993 Jul;54(1):23-7. doi: 10.1038/clpt.1993.104. PMID 8330461
- [Result] Hyvonen T, Keinanen TA, Khomutov AR, Khomutov RM, Eloranta TO. Monitoring of the uptake and metabolism of aminooxy analogues of polyamines in cultured cells by high-performance liquid chromatography. J Chromatogr. 1992 Feb 7;574(1):17-21. doi: 10.1016/0378-4347(92)80093-6. PMID 1629283
- [Result] Lou G, Zhang M, Minuk GY. Effects of acute ethanol exposure on polyamine and gamma-aminobutyric acid metabolism in the regenerating liver. Alcohol. 1999 Nov;19(3):219-27. doi: 10.1016/s0741-8329(99)00050-6. PMID 10580511